CLINICAL TRIAL: NCT04825314
Title: Noble Metal Alloy Coated Versus Silicone Foley Catheter in Patients With Long Term Catheterization: A Prospective Randomized Controlled Study
Brief Title: Noble Meta Alloy Coated Catheters in Patients With Long Term Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Tamer Abou Youssif, Associate Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0106462
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Urinary Tract Infections; Catheter Infection; Catheter-Related Infections; Infection
Keywords: catheter; UTI; Foley catheter; Nobel Metal Alloy catheter
MeSH Terms: conditions — Urinary Tract Infections; Catheter-Related Infections; Infections | interventions — Urinary Catheters

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bactiguard urethral catheter (Active Comparator): Group A: Fifty Patients with urethral catheter using noble metal alloy coated catheter (Bactiguard AB, Stockholm ,Sweden).
  Interventions: Device: Urethral catheter
- Silicone Foley urethral catheter (Active Comparator): Group B: Fifty Patients with urethral catheter using silicone Foley catheter (Well Lead, Guangzhou, China).
  Interventions: Device: Urethral catheter

INTERVENTIONS:
Device: Urethral catheter — All Patients will have urethral catheterization with either Noble Metal Alloy coated catheter or Silicon Foley catheter.

SUMMARY:
Eighty percent of nosocomial UTI caused by indwelling urinary catheters and so known-as catheter-associated UTI. CAUTI leads to multiple local and systemic derangements such as suprapubic pain, dysuria, cystitis, pyelonephritis, septicemia, and even septic shock.

This study will be conducted up on 100 patients (50 per each group) with long term catheterization to assess efficacy of noble metal alloy coated catheter in reducing CAUTI.

DETAILED DESCRIPTION:
This prospective controlled randomized study conducted upon 100 patients at Alexandria University hospital from 21 May 2020 to 21 December 2020. Patients enrolled will be divided into two equal groups according to the urethral catheter inserted

The institutional ethics committee for research approved the study. Written informed consent was obtained from all participants. In addition to taking the patients' medical history and completing general and physical examinations, physicians will choose proper catheter size all perform catheterization using aseptic technique according to guidelines of proper aseptic catheterization. Urologist ensures comparable catheter size and amount of balloon inflation.

An aseptic non-touch technique (ANTT) must be used to obtain catheter specimen urine following these steps:

* After catheterization apply clamp 10 cm distal to meatus then after few minutes clean the drainage port with alcohol and allow to dry then insert the syringe tip into the drainage port.
* Three to five ml of urine collected in sterile disposable plastic cup at day zero (within 2 hours of catheterization), day ten and day twenty post catheterization.
* The urine subjected to routine urine analysis, urine culture and sensitivity.

Appropriate statistical tests will be used to indicate the frequency and type of CAUTI as well as to assess catheter tolerance in each arm, followed by a comparison to conclude the results.

ELIGIBILITY:
Inclusion Criteria:

- Patient under age of 80 years old who need prolonged urethral catheterization (more than 2 weeks) as a method of bladder drainage.

Exclusion Criteria:

* Patients with current or recent symptomatic urinary tract infection.
* Antibiotic use currently or within 7 days prior to inclusion.
* Known hypersensitivity to latex, silver salts or hydrogel.
* Patients with recent surgical intervention in the urinary tract.
* Patients with anatomic or functional upper urinary tract issues (e.g reflux, stones, etc.)
* Uncontrolled DM. Patients on corticosteroid treatment. Immunosuppressed patients. Patients received pelvic irradiation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-05-21 (Estimated); Study Completion 2021-06-21 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infection | 14 days
  incidence of culture documented symotomatic urinary tract infection

SECONDARY OUTCOMES:
Catheter tolerance | 14 days
  Catheter tolerance looks for discomfort or pain. Discomfort is an uncomfortable sensation due to the presence of a foreign object in the urethra without pain. The presence of actual pain is measured using VAS scoring system from zero to ten, so that a zero means no pain and a tenth means very severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aljohi AA, Hassan HE, Gupta RK. The efficacy of noble metal alloy urinary catheters in reducing catheter-associated urinary tract infection. Urol Ann. 2016 Oct-Dec;8(4):423-429. doi: 10.4103/0974-7796.192099. PMID 28057985